CLINICAL TRIAL: NCT02609087
Title: Comparison the Effect on Cerebral Oxygenation by Sevoflurane-remifentanil or Propofol-remifentanil Anesthesia Using Near-infrared Spectroscopy in Patients Undergoing Carotid Endarterectomy)
Brief Title: Effect on Cerebral Oxygenation by Sevoflurane or Propofol Using Near-infrared Spectroscopy in Carotid Endarterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Seongtae Jeong, Associated professor, Anesthesiolgoy and Pain Medicine, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2015-159
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Experimental): adjust the end-tidal sevoflurane (sevofran inhaler, Hana pharmacy, Korea) concentration maintaining the 40 ~ 50 BIS (bispectral index) with 3 ng/ml of remifentanil using TCI (target controlled infusion) pump
  Interventions: Drug: Sevoflurane
- Propofol (Experimental): adjust propofol (FRESOFOL MCT INJ 2% (vial), Fresinus Kabi Korea) concentration maintaining the 40 ~ 50 BIS (bispectral index) with 3 ng/ml of remifentanil using TCI (target controlled infusion) pump
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane
  Arms: Sevoflurane
Drug: Propofol
  Arms: Propofol

SUMMARY:
The aim of this study is comparing the effect on cerebral oxygenation by sevoflurane-remifentanil or propofol-remifentanil anesthesia in patient undergoing carotid endarterectomy. Cerebral oxygenation is measured by near-infrared spectroscopy. Sevoflurane and propofol reduce the cerebral metabolic rate for oxygen in similar degree. Propofol decrease the cerebral blood flow by dose-dependent manner, however, sevoflurane increase the cerebral blood flow in the concentration of avobe 1 MAC. Both drugs are widely used in general anesthesia for neurosurgical procedure, and their effect on cerebral oxygenation are acceptable. There is little data about the effect of general anethetics on cerebral oxygenation in patients undergoing carotid endarterectomy, who have imparied cerebral circulation. Our hypothesis is sevoflurane will show better cerebral oxygenation than propofol in patient have impaired cerebral circulation.

DETAILED DESCRIPTION:
This study is performed by monitoring the cerebral oxygenation using near-infrared spectroscopy from general anesthesia induction to 10 min after releasing the carotid artery clipping.

Study group: Sevoflurane - remifentanil anesthesia group (S) Propofol - remifentanil anesthesia group (R)

Monitoring: near-infrared spectroscopy (SOMA sensor) BIS, HR, arterial blood pressure, SpO2, body temperature

Patient seletion

* inclusion criteria

  * American Society of Anesthesiologist (ASA) physical status 1-3
  * 18 ~ 70 years
  * patient who agree with informed concent
* exclusion criteria

  * ASA physical status > 4
  * preoperative SpO2 < 97%
  * patient who has other neurologic disease not related to carotid endarterectomy

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status 1-3
* 18 ~ 70 years
* patient who agree with informed consent

Exclusion Criteria:

* ASA physical status > 4
* preoperative SpO2 < 97%
* patient who has other neurologic disease not related to carotid endarterectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
cerebral oxygenation measured by near-infrared spectroscopy | one year

CONTACTS AND LOCATIONS:
Overall Officials: Seongtae Jeong, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

REFERENCES:
- [Derived] Park S, Yook K, Yoo KY, Choi JI, Bae HB, You Y, Jin B, Jeong S. Comparison of the effect of sevoflurane or propofol anesthesia on the regional cerebral oxygen saturation in patients undergoing carotid endarterectomy: a prospective, randomized controlled study. BMC Anesthesiol. 2019 Aug 17;19(1):157. doi: 10.1186/s12871-019-0820-9. PMID 31421685